CLINICAL TRIAL: NCT05936450
Title: Assessment Of Healing After Periodontal Flap Surgery Using Periostin Levels In Gingival Crevicular Fluid With And Without The Use Of Placental Extracts
Brief Title: Assessment Of Healing After Periodontal Flap Surgery With And Without The Use Of Placental Extracts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Prabhuji MLV (Other)
Responsible Party: Sponsor-Investigator, Dr Prabhuji MLV, Professor, Head of Department, Krishnadevaraya College of Dental Sciences & Hospital
Organization: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_112276
Record Dates: First submitted 2023-02-06; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Periodontal Diseases; Periodontal Pocket; Periodontitis
Keywords: placental extract; periostin; healing
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Experimental): placentrex gel + Open Flap Debridement
  Interventions: Biological: delivery of placentrex gel after open flap debridement; Procedure: Open Flap Debridement
- control group (Active Comparator): Open Flap Debridement alone
  Interventions: Procedure: Open Flap Debridement

INTERVENTIONS:
Biological: delivery of placentrex gel after open flap debridement — placentrex gel is placed after open flap debridement only in the test group
  Arms: test group
Procedure: Open Flap Debridement — Open Flap Debridement done in both test and control groups

SUMMARY:
All 16 chronic periodontitis (CP) subjects were clinically examined regarding the following clinical periodontal parameters: plaque index (PI), gingival index (GI), bleeding index (BI), Pocket Probing Depth (PPD) and Relative Attachment Loss (RAL) which were recorded for all patients at baseline and 3 months after surgical periodontal treatment.

Pre- surgical procedure:

After the clinical parameters were recorded, Phase I therapy (full mouth scaling, root planning and oral hygiene instructions) was carried out.

The patients were then put under observation to assess the oral hygiene practice and the response of the gingival tissue to Phase I therapy.

After two weeks, patients were recalled and based on further treatment protocol, periodontal flap surgery was planned. Group A (Test Group) underwent periodontal flap surgery during which placental extract was applied. Group B (Control Group) underwent periodontal flap surgery alone.

Surgical procedure The operative sites were anaesthetized with 2% lignocaine hydrochloride with adrenaline (1:180000).

Crevicular incisions were made using Bard Parker No.15 blade on the facial and lingual/palatal surface of each tooth segment or area involved.

A full thickness mucoperiosteal flap was reflected using periosteal elevator taking care to preserve the maximum amount of tissue in the flap. After exposure the granulation tissue was removed, the root surfaces were planed and the flap was trimmed of tissue tags to facilitate healing.

The flap was approximated using interrupted sutures (mersilk 3-0) and a periodontal dressing was placed above it.

Local delivery of the placental extract In group A patients (test group) after open flap debridement 1ml of human placental extracts gel (Placentrex - the original research product of Albert David Limited, India, a drug obtained from fresh term healthy human placentae) was dispensed in a dappen dish.

Gelatin foam (Abgel, Sri Gopal Krishna Labs, Pvt.Ltd. India) was cut into small beads of 1 sq.mm and allowed to soak in the placental gel for a few seconds. These gelatin beads soaked in gel are placed into the surgical site locally with the help of a graft carrier and condensed into the defect area.

To prevent uncontrolled spill-over effects of the gel, mild pressure was applied over the flap with the wet gauze and excess gel was removed and Coe Pak was placed.

While in group B(control group), after open flap debridement, this step is omitted.

Post-operative care Antibiotics and analgesics are prescribed two times a day for five days. Patients were instructed to refrain from chewing hard or sticky foods, brushing near the treated areas or using any interdental aids for 1 week.

The use of mouthwash was avoided during the observation period. All patients were placed on a strict maintenance schedule following surgery. The sutures were removed 10 days later.

Recall appointments were scheduled once in 10 days for the 1st month. At every recall appointment, oral hygiene was checked.

At 3rd month, the clinical parameters were recorded in both the groups. The difference between pre and post-operative values was assessed and then statistically analysed

DETAILED DESCRIPTION:
All 16 chronic periodontitis (CP) subjects were clinically examined regarding the following clinical periodontal parameters: plaque index (PI), gingival index (GI), bleeding index (BI), Pocket Probing Depth (PPD) and Relative Attachment Loss (RAL) which were recorded for all patients at baseline and 3 months after surgical periodontal treatment.

Technique to ascertain the Probing Pocket Depth (PPD) and Relative attachment Level (RAL) at the treatment sites: A customized acrylic stent was fabricated for each patient for providing a reproducible insertion axis for the probe. The stent was grooved in an occluso-apical direction for the above mentioned purpose. The following clinical parameters were recorded with the help of a Hu Friedy UNC 15 probe.

Measurements were taken from stent to deepest probing depth to record Probing pocket depth (PPD) while Relative Attachment level (RAL) were recorded by subtracting the length of deepest probing depth from stent by the length from stent to cemento-enamel junction.

Collection of Gingival Crevicular Fluid(GCF) GCF samples were obtained from the buccal aspects of the selected site. The sites were isolated by cotton rolls, rinsed with water and dried with a gentle air spray directed perpendicular to the gingival margin.

Removal of supra-gingival plaque was completed utilizing dry gauze, and a sterile filter paper strip((ORAFLOW). ® was gently inserted into the entrance of the selected site until the first sign of resistance was felt for 30 sec. Samples contaminated with gingival bleeding were excluded.

The GCF sample volume will be measured in a calibrated appliance (Periotron 8000 Proflow Inc., Amityville, NY, USA) TM, after which the reading will be converted to an actual volume (µl) by reference to the standard curve.

The strips from the selected site will be transferred in micro centrifuged tubes containing 100(µl) of phosphate buffer saline.

The samples will be stored at -80 0C till the assay is performed using Enzyme Linked Immuno Sorbent Assay (ELISA) kit obtained from (GENXBIO)TM, as per the manufacturer's instructions.

The same steps are repeated at baseline, 6 weeks and 3 months.

Pre- surgical procedure:

After the clinical parameters were recorded, Phase I therapy (full mouth scaling, root planning and oral hygiene instructions) was carried out.

The patients were then put under observation to assess the oral hygiene practice and the response of the gingival tissue to Phase I therapy.

After two weeks, patients were recalled and based on further treatment protocol, periodontal flap surgery was planned. Group A (Test Group) underwent periodontal flap surgery during which placental extract was applied. Group B (Control Group) underwent periodontal flap surgery alone.

Surgical procedure The operative sites were anaesthetized with 2% lignocaine hydrochloride with adrenaline (1:180000).

Crevicular incisions were made using Bard Parker No.15 blade on the facial and lingual/palatal surface of each tooth segment or area involved.

A full thickness mucoperiosteal flap was reflected using periosteal elevator taking care to preserve the maximum amount of tissue in the flap. After exposure the granulation tissue was removed, the root surfaces were planed and the flap was trimmed of tissue tags to facilitate healing The flap was approximated using interrupted sutures (mersilk 3-0) and a periodontal dressing was placed above it.

Local delivery of the placental extract In group A patients (test group) after open flap debridement 1 ml of human placental extracts gel (Placentrex - the original research product of Albert David Limited, India, a drug obtained from fresh term healthy human placentae) was dispensed in a dappen dish.

Gelatin foam (Abgel, Sri Gopal Krishna Labs, Pvt.Ltd. India) was cut into small beads of 1 sq.mm and allowed to soak in the placental gel for a few seconds. These gelatin beads soaked in gel are placed into the surgical site locally with the help of a graft carrier and condensed into the defect area.

To prevent uncontrolled spill-over effects of the gel, mild pressure was applied over the flap with the wet gauze and excess gel was removed and Coe Pak was placed.

While in group B(control group), after open flap debridement, this step is omitted.

Post-operative care Antibiotics and analgesics are prescribed two times a day for five days. Patients were instructed to refrain from chewing hard or sticky foods, brushing near the treated areas, or using any interdental aids for 1 week.

The use of mouthwash was avoided during the observation period. All patients were placed on a strict maintenance schedule following surgery. The sutures were removed 10 days later.

Recall appointments were scheduled once in 10 days for the 1st month. At every recall appointment, oral hygiene was checked.

At 3rd month, the clinical parameters were recorded in both the groups. The difference between pre and post-operative values was assessed and then statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age group of 25 to 55 years.
2. Patients with chronic periodontitis, with probing pocket depth (PPD) ≥ 6mm and presence of alveolar defect.
3. Systemically healthy subjects.
4. Patients who are compliant.
5. Patients who had not received any periodontal treatment in the last six months and anti-microbial therapy in past three months.

Exclusion Criteria:

1. Pregnant and Lactating females.
2. Aggressive periodontitis.
3. Presence of pulpal or periapical involvement.
4. Patients with known conditions precluding any elective surgery.
5. Smokers.
6. Teeth with poor prognosis.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Pocket Probing Depth (PPD) | Change from Baseline Periodontal disease at 3 months
  Measurements were taken from stent to deepest probing depth to record Probing pocket depth (PPD)
Relative Attachment Loss (RAL) | Change from Baseline Periodontal disease at 3 months
  Relative Attachment level (RAL) were recorded by subtracting the length of deepest probing depth from stent by the length from stent to cemento-enamel junction.
Plaque Index (PI) | Change from Baseline Periodontal disease at 3 months
  The scoring is done on the entire dentition or on selected teeth. Plaque of the cervical third of the tooth is evaluated with no attention to plaque that has extended to the middle or incisal thirds. The surfaces examined are the four gingival areas of the tooth i.e. the disto-facial, facial, mesio-facial, and lingual surfaces.
  Scoring criteria:
  0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be in situ only after application of disclosing solution or by using probe on the tooth surface.
  2. Moderate accumulation of soft deposit within the gingival pocket, or the tooth and the gingival margin which can be seen with naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Gingival Index (GI) | Change from Baseline Periodontal disease at 3 months
  The severity of gingivitis is scored on the mesiofacial and distofacial papillae, facial and lingual margin of selected teeth.A blunt instrument is used to assess the bleeding potential of tissues.The index relies entirely on visual criteria of gingivitis and eliminates the use of probing or pressure to establish the presence or absence of bleeding.
  Score Criteria 0 Absence of inflammation/normal gingiva
  1. Mild inflammation, slight change in color, slight edema; no bleeding on probing
  2. Moderate inflammation; moderate glazing, redness, edema and hypertrophy. Bleeding on probing.
  3. Severe inflammation; marked redness, hypertrophy and ulceration. Tendency to spontaneous bleeding
     * G.I SCORE = Total score / No of teeth examined
  Rating Score Mild gingivitis=0.1-1.0 Moderate gingivitis=1.1-2.0 Severe gingivitis =2.1-3.0
Bleeding Index (BI) | Change from Baseline Periodontal disease at 3 months
  The gingival bleeding index of Ainamo J and Bay I was developed as an easy and suitable way for assessing a patient's progress in Plaque control. The presence or absence of gingival bleeding is determined by gentle probing of the gingival crevice with a periodontal probe. The appearance of bleeding within 10 seconds indicates a positive score, which is expressed as percentage of the total number of gingival margin examined.
  • Scoring criteria: Score Criteria 0 No bleeding present on probing within 10 seconds
  1 Bleeding present on probing within 10 seconds.
  • Calculation : = Total score / No of teeth examined
periostin levels | Change from Baseline Periodontal disease at 3 months
  Collection of gingival crevicular fluid GCF samples were obtained from the buccal aspects of the selected site. The sites were isolated by cotton rolls, rinsed with water and dried with a gentle air spray directed perpendicular to the gingival margin.
  Removal of supra-gingival plaque was completed utilizing dry gauze, and a sterile filter paper strip((ORAFLOW). ® was gently inserted into the entrance of the selected site until the first sign of resistance was felt for 30 sec. Samples contaminated with gingival bleeding were excluded.
  The GCF sample volume will be measured in a calibrated appliance (Periotron 8000 Proflow Inc., Amityville, NY, USA) TM, after which the reading will be converted to an actual volume (µl) by reference to the standard curve.

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

REFERENCES:
- [Background] Padial-Molina M, Volk SL, Rios HF. Preliminary insight into the periostin leverage during periodontal tissue healing. J Clin Periodontol. 2015 Aug;42(8):764-772. doi: 10.1111/jcpe.12432. Epub 2015 Aug 19. PMID 26202398
- [Background] Sharma A, Sharma S, Nagar A. Comparative Evaluation to Assess the Effect of SRP With or Without Human Placental Extracts as Local Drug Delivery in Treatment of Localized Periodontal Pocket-A Randomized Controlled Clinical Trial.